CLINICAL TRIAL: NCT05678218
Title: Preoperative Evaluation of Lymph Nodes of Cholangiocarcinoma - a Registration Study
Brief Title: Preoperative Evaluation of Lymph Nodes of Cholangiocarcinoma
Acronym: POELH-II
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Dr. L.M.J.W. (Lydi) van Driel, Gastroenterologist, MD, PhD, Erasmus Medical Center
Other Study IDs: MEC-2022-0402
Record Dates: First submitted 2022-12-23; First posted 2023-01-10 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Hilar Cholangiocarcinoma; Intrahepatic Cholangiocarcinoma; Common Bile Duct Neoplasms; Cholangiocarcinoma; Adenocarcinoma
Keywords: Endoscopic Ultrasound; Fine Needle Aspiration; Fine Needle Biopsy; Lymph Node; Adenocarcinoma
MeSH Terms: conditions — Klatskin Tumor; Cholangiocarcinoma; Common Bile Duct Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Presumed resectable perihilar, intrahepatic or mid-common bile duct (CBD) cholangiocarcinoma
  Interventions: Procedure: Endoscopic Ultrasound registration

INTERVENTIONS:
Procedure: Endoscopic Ultrasound registration — Registration of all findings during Endoscopic Ultrasound

SUMMARY:
The goal of this observational cohort study is to assess the yield of preoperative endoscopic ultrasound focussed on lymph nodes in patients with presumed resectable perihilar (pCCA), intrahepatic (iCCA) or mid-common bile duct (CBD) cholangiocarcinoma. The main questions it aims to answer is:

1. The number of patients precluded from surgical work-up due to positive regional or extraregional lymph nodes identified by endoscopic ultrasound guided tissue acquisition
2. Characteristics during endoscopic ultrasound of lymph nodes associated with malignancy

ELIGIBILITY:
Inclusion Criteria:

* Presumed resectable pCCA OR
* Presumed resectable iCCA OR
* Presumed resectable mid-common bile duct CCA OR
* Presumed unresectable pCCA worked-up for Liver Transplantation AND
* Written informed consent must be given according to International Council on Harmonisation/Good Clinical Practice guidelines, and national/local regulations AND
* Age > 18 years.

Exclusion Criteria:

* Patients with a history of treated CCA
* Patients with CCA for which a pancreatoduodenectomy is indicated, based on cross-sectional imaging
* Patients with a history of treated liver malignancy
* Patients with a contra-indication for EUS-tissue acquisition (f.e. uncorrectable coagulopathy or platelet disorder), in line with current clinical practice

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected iCCA or pCCA who have a presumed resectable carcinoma will be invited to participate. Patients with CCA distal from the cystic junction but proximal from the pancreatic body are eligible for inclusions as well, as treatment is similar to Bismuth I pCCA. In other words, all patients with CCA that is not distal CCA for which a pancreato-duodenectomy is indicated, are eligible for inclusion. Also patients with presumed unresectable pCCA who are worked-up for liver transplantation are invited to participate. At time of inclusion a definitive diagnosis of iCCA/pCCA is not obligatory, since definitive diagnosis of CCA is sometimes confirmed during the preoperative EUS through EUS guided biopsy of the mass. The probable diagnosis of iCCA/pCCA and the suspected resectability will be established during the multidisciplinary meeting, based on clinical symptoms, cross-sectional imaging, endoscopy and laboratory tests.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Lymph nodes identified compared to imaging | Through study completion, max 1 year
  Number of lymph nodes correctly identified based on visualization and biopsy in comparison to cross-sectional imaging
Lymph nodes identified compared to surgery | Through study completion, max 1 year
  Number of lymph nodes correctly identified based on visualization and biopsy in comparison to surgery, in the patients in which this is performed

SECONDARY OUTCOMES:
Endoscopic Ultrasound (EUS)-characteristics predictive for malignant involvement of lymph nodes | Through study completion, max 1 year
  Rate of malignant lymph nodes in which a certain characteristic is present (f.e. shape of the lymph node), in comparison to benign lymph nodes.
Different locations of positive lymph nodes and its effect on survival | Through study completion, max 1 year
  Days of survival after EUS and surgery, stratified per cholangiocarcinoma type, as well as lymph node locations
Short term and long term complications of the EUS (+/- tissue acquisition) procedure for patients with pCCA and iCCA | Through study completion, max 1 year
  Short term (<30 days)
  * Sedation related: consisting of cardiovascular-related complications (cardiac arrhythmias, myocardial ischemia/infarction), respiratory- related complications (respiratory depression, hypoxia, airway obstruction, pulmonary aspiration of gastric contents) and allergic reactions.
  * Hemorrhage (outside peritoneal wall): defined as clinical evidence of bleeding with a hemoglobin drop of >3g/dl with the need for resuscitation or additional intervention
  * Perforation: defined as evidence of air or luminal contents outside the gastro-intestinal tract together with clinical symptoms, requiring percutaneous drainage or surgery
  * Mortality
  Long term (>30 days)
  - Tumor seeding; defined as proof of carcinoma in the biopsy tract during follow-up or at autopsy

CONTACTS AND LOCATIONS:
Locations (7):
- University Hospital of Ghent, Ghent, Belgium
- Netherlands (6):
  - Maastricht UMC+, Maastricht, Limburg
  - Amsterdam University Medical Center, Amsterdam, North Holland
  - University Medical Center Groningen, Groningen, Provincie Groningen
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus University Medical Center, Rotterdam, South Holland
  - University Medical Center Utrecht, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] de Jong DM, Lammers WJ, van Driel LMJW. Time to standardize preoperative EUS for lymph node staging in resectable extrahepatic cholangiocarcinoma. J Hepatol. 2025 Dec;83(6):e290-e291. doi: 10.1016/j.jhep.2025.06.031. Epub 2025 Jul 9. No abstract available. PMID 40645595
- [Background] de Jong DM, van de Vondervoort S, Dwarkasing RS, Thomeer MGJ, Doukas M, Voermans RP, Verdonk RC, Polak WG, de Jonge J, Bruno MJ, Van Driel LMJW, Groot Koerkamp B. Endoscopic ultrasound with tissue acquisition of lymph nodes in patients with potentially resectable intrahepatic cholangiocarcinoma. Endosc Int Open. 2024 Aug 23;12(8):E998-E1005. doi: 10.1055/a-2366-2592. eCollection 2024 Aug. PMID 39184062
- [Background] Malikowski T, Levy MJ, Gleeson FC, Storm AC, Vargas EJ, Topazian MD, Abu Dayyeh BK, Iyer PG, Rajan E, Gores GJ, Roberts LR, Chandrasekhara V. Endoscopic Ultrasound/Fine Needle Aspiration Is Effective for Lymph Node Staging in Patients With Cholangiocarcinoma. Hepatology. 2020 Sep;72(3):940-948. doi: 10.1002/hep.31077. Epub 2020 Jul 9. PMID 31860935
- [Background] Gleeson FC, Rajan E, Levy MJ, Clain JE, Topazian MD, Harewood GC, Papachristou GI, Takahashi N, Rosen CB, Gores GJ. EUS-guided FNA of regional lymph nodes in patients with unresectable hilar cholangiocarcinoma. Gastrointest Endosc. 2008 Mar;67(3):438-43. doi: 10.1016/j.gie.2007.07.018. Epub 2007 Dec 3. PMID 18061597
- [Background] Larghi A, Rimbas M, Ardito F, Rizzatti G, Giuliante F. Letter to the Editor: EUS-FNA for Lymph Nodes Staging in Cholangiocarcinoma: Should It Become Standard of Care? Hepatology. 2020 Oct;72(4):1496. doi: 10.1002/hep.31266. No abstract available. PMID 32277489
- [Background] de Jong DM, van de Vondervoort S, Dwarkasing RS, Doukas M, Voermans RP, Verdonk RC, Polak WG, de Jonge J, Koerkamp BG, Bruno MJ, van Driel LMJW. Endoscopic ultrasound in patients with resectable perihilar cholangiocarcinoma: impact on clinical decision-making. Endosc Int Open. 2023 Feb 2;11(2):E162-E168. doi: 10.1055/a-2005-3679. eCollection 2023 Feb. PMID 36741342
- [Background] de Jong DM, den Hoed CM, Willemssen FEJA, Thomeer MGJ, Bruno MJ, Koerkamp BG, de Jonge J, Alwayn IPJ, van Hooft JE, Hoogwater F, van der Heide F, Inderson A, van Vilsteren FGI, van Driel LMJW. Impact of EUS in liver transplantation workup for patients with unresectable perihilar cholangiocarcinoma. Gastrointest Endosc. 2024 Apr;99(4):548-556. doi: 10.1016/j.gie.2023.10.047. Epub 2023 Oct 27. PMID 37890597
- See also: Related Info — https://onderzoekmetmensen.nl/en/trial/49893